CLINICAL TRIAL: NCT04905368
Title: Tolerability of a Topical Dermo-cosmetic Product in Acne-prone Subjects
Brief Title: Safety Evaluation of SS-POR11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klynical Consulting & Services (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SS-POR11
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SS-POR11 — Topical composition containing probiotic strains derived from human skin (SS-POR11). Participants will be instructed to apply it topically to face, twice weekly for the duration of the trial.

SUMMARY:
The goal of the present study is to assess the safety of a topical probiotic (probiotic strain; SS-POR11) on acne prone-skin, and the impact of SS-POR11 on the distribution of porphyrins, in subjects with mild-to-moderate acne [Investigator's Global Assessment (IGA) 1-3].

ELIGIBILITY:
Inclusion Criteria:

* Participant's first language of French or English, given the written language of the ICF
* Participants willing to sign the ICF upon entering the study
* Participant must be willing and able (in the PI's opinion) to comply with all study requirements
* Participant must be aged 18-40 years
* Participant must have a screening and baseline IGA score of 1 (rare blemishes/clear skin) or 2-3 (mild to moderate facial acne vulgaris)
* Participant must agree to appear on all evaluation days and conform to all study-related instructions
* Participant must agree not to undergo any topical treatments in the areas under investigation during the study period

Exclusion Criteria:

* Participants under the age of 18 years or over the age of 40
* Refusal to sign the ICF
* Participants has any injuries or tumors in the areas under investigation
* Participant has a recent (i.e., 3 months) surgery or invasive treatment in the areas under investigation
* Use of oral antibiotics within 4 weeks prior to start of study
* Use of oral or topical "probiotic" products within one month prior to start of study
* Prior (3 months) or planned use of chemical peels, microdermabrasion, microneedling, or exfoliants during the course of the study
* Participant is using or has used within 3 months drugs such as corticosteroids, immunosuppressants, or others collagen-production inhibitors
* Participant is pregnant or lactating or wishes to get pregnant within the next 3 months, or refuses to use appropriate contraceptive method (in case of women of childbearing potential)
* Participant has active herpes simplex in the investigated areas or a history of herpes labialis with four or more outbreaks in the 12 months prior to baseline
* Participant has immunocompromising diseases; any known allergy or hypersensitivity to any of the ingredients of the investigational product
* Participants possessing any of the contraindications for use of SS-POR11
* Participant has tattoos, piercings, excessive scarring (e.g., hypertrophic or keloid scars) in the areas under investigation
* Current or prior (3 months) change in the use of retinoids; Initiated use of hormones or change in dose of hormonal replacement therapy within 3 months; and any other criteria that at the discretion of the Investigator, could interfere with study assessments or expose the subject to undue risk by study participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and Serious AEs (SAEs) associated with the topical use of SS-POR11 | Baseline
  Frequency of AEs and SAEs
Signs of intolerance associated with the topical use of SS-POR11 | Week 2
  Frequency of signs of intolerance, via evaluation of the Skin Tolerability Test
Subject sensitivity to SS-POR11 | Baseline
  Frequency of signs of sensitivity, via evaluation of the Skin Tolerability Test.
Adverse events (AEs) and Serious AEs (SAEs) associated with the topical use of SS-POR11 | Week 2
  Frequency of AEs and SAEs
Adverse events (AEs) and Serious AEs (SAEs) associated with the topical use of SS-POR11 | Week 4
  Frequency of AEs and SAEs
Signs of intolerance associated with the topical use of SS-POR11 | Week 4
  Frequency of signs of intolerance, via evaluation of the Skin Tolerability Test

SECONDARY OUTCOMES:
Porphyrin distribution | Week 2, Week 4
  Efficacy of SS-POR11 to reduce levels of porphyrins on the skin, as assessed by the VISIA® Skin Analysis System.
  Average percent change in facial porphyrin distribution
Investigator Global Assessment (IGA) | Week 2, Week 4
  Frequency of subjects displaying at least a one-point improvement on the IGA, at follow up visits compared to baseline. The IGA is an ordinal scale with five grades corresponding to increasing severities of acne (e.g., 0 to 4).

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlyn Enright, Study Director — Klynical Consulting & Services
Locations (1):
- Klynical Consulting & Services, Westmount, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No